CLINICAL TRIAL: NCT02364674
Title: Transplant Optimization Using Functional Imaging
Acronym: TROFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FLUIDDA nv (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FLUI-2014-103_USA
Record Dates: First submitted 2015-02-05; First posted 2015-02-18 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2016-02

CONDITIONS: Bronchiolitis Obliterans; Lung Transplant Rejection
Keywords: HRCT; High Resolution Computed Tomography scans; Functional Respiratory Imaging; FRI; Computed Tomography; CT; Bronchiolitis Obliterans; BOS; Lung Transplant
MeSH Terms: conditions — Bronchiolitis Obliterans

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HRCT scans (Experimental): HRCT scan will be taken
  Interventions: Radiation: High Resolution Computed Tomography scan

INTERVENTIONS:
Radiation: High Resolution Computed Tomography scan — a HRCT scan at Functional Residual Capacity (FRC) and Total Lung Capacity (TLC) will be taken on visit 1, visit 2, visit 3, visit 4 and visit 5.
  An Upper Airway (UA) scan will be taken on visit 1.
  Other Names: HRCT scan

SUMMARY:
The objective of this study is to detect Bronchiolitis Obliterans Syndrome (BOS) in an early stage using the outcome parameters generated by Functional Respiratory Imaging (FRI). Robust and automated segmentation algorithms will be developed for these parameters, focusing on quantitative computed tomography (CT) image analyses to provide the physician a more sensitive diagnostics tool. The evolution of BOS over time will be monitored using non-rigid image registration methods.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient ≥ 18 years old
* Written informed consent obtained
* Patient who had undergone a lung transplant a year ago or more.
* Female patient of childbearing potential who confirm that a contraception method was used at least 14 days before visit 1 and will continue to use a contraception method during the study
* The patient must be able to perform the lung monitoring at home.

Exclusion Criteria:

* Pregnant or lactating female
* Known history of or active airways or anastomotic complications requiring intervention such as stenting or dilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-02; Primary Completion 2017-01-09 (Actual); Study Completion 2017-01-09 (Actual)

PRIMARY OUTCOMES:
Airway Volume (iVaw) | 12 months
  Exploratory imaging endpoints: HRCT-scan will be taken at visit 1 - visit 5.
Airway Resistance (iRaw) | 12 months
  Exploratory imaging endpoints: HRCT-scan will be taken at visit 1 - visit 5.
Specific Airway Volume (siVaw) | 12 months
  Exploratory imaging endpoints: HRCT-scan will be taken at visit 1 - visit 5.
Specific Airway Resistance (siRaw) | 12 months
  Exploratory imaging endpoints: HRCT-scan will be taken at visit 1 - visit 5.
Lobe volumes (iVlobes) | 12 months
  Exploratory imaging endpoints: HRCT-scan will be taken at visit 1 - visit 5.
Air trapping | 12 months
  Exploratory imaging endpoints: HRCT-scan will be taken at visit 1 - visit 5.
Internal Lobar Airflow Distribution | 12 months
  Exploratory imaging endpoints: HRCT-scan will be taken at visit 1 - visit 5.
Low Attenuation or Emphysema Score | 12 months
  Exploratory imaging endpoints: HRCT-scan will be taken at visit 1 - visit 5.
Blood Vessel Density or Fibrosis Score | 12 months
  Exploratory imaging endpoints: HRCT-scan will be taken at visit 1 - visit 5.
Airway Wall Thickness | 12 months
  Exploratory imaging endpoints: HRCT-scan will be taken at visit 1 - visit 5.

CONTACTS AND LOCATIONS:
Overall Officials: David Lederer, M.D., M.S., Principal Investigator — Columbia University; James Lee, M.D., M.S., Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Columbia University Medical Center, New York, New York
  - Hospital of the University of Pennsylvania, Gibson, Pennsylvania